CLINICAL TRIAL: NCT02649751
Title: A Phase II, Dose Ranging, Multicenter, Double-blind, Placebo Controlled Study to Evaluate Safety and Effects of (R)-Roscovitine in Adults Subjects With Cystic Fibrosis, Carrying 2 Cystic Fibrosis Causing Mutations With at Least One F508del-CFTR Mutation and Chronically Infected With Pseudomonas Aeruginosa, a Study Involving 36 CF Patients (24 Treated, 12 Controls). ROSCO-CF.
Brief Title: Evaluation of (R)-Roscovitine Safety and Effects in Subjects With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation
Acronym: ROSCO-CF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The centers have no longer patients. In September 2018, set up of a competitive international study.
Sponsor: University Hospital, Brest (Other)
Collaborators: ManRos Therapeutics (Unknown); Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RB 15.098 (ROSCO CF)
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2018-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Roscovitine; Seliciclib; CYC202
MeSH Terms: conditions — Cystic Fibrosis | interventions — Roscovitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): 200 mg roscovitine (8) or placebo (4) once daily for 4 cycles of 7 days (4 days "on" and 3 days "off")
  Interventions: Drug: Roscovitine; Drug: Placebo
- Group 2 (Experimental): 400 mg roscovitine (8) or placebo (4) once daily for 4 cycles of 7 days (4 days "on" and 3 days "off")
  Interventions: Drug: Roscovitine; Drug: Placebo
- Group 3 (Experimental): 400 mg roscovitine (8) or (4) placebo twice daily for cycles of 7 days (4 days "on" and 3 days "off")
  Interventions: Drug: Roscovitine; Drug: Placebo

INTERVENTIONS:
Drug: Roscovitine — Roscovitine is an experimental drug candidate in the family of pharmacological cyclin-dependent kinase (CDK) inhibitors that preferentially inhibit multiple enzyme targets including CDK2, CDK7 and CDK9. Seliciclib is a 2,6,9-substituted purine analog.
  Other Names: Seliciclib; CYC202
Drug: Placebo — The placebo treatment is lactose capsule.

SUMMARY:
This is a phase II, dose ranging, multicenter, randomized, double-blind, placebo-controlled study.

The aim of this study is to assess the safety of increasing doses of roscovitine administered orally for 4 cycles of 4 consecutive days (treatment "on") separated by a 3 days treatment free period (treatment "off") in adult CF subjects with Cystic Fibrosis carrying 2 Cystic Fibrosis causing mutations with at least one F508del-CFTR mutation and chronically infected with Pseudomonas aeruginosa.

This study involved 36 Cystic Fibrosis patients: 24 treated and 12 controls.

DETAILED DESCRIPTION:
ROSCO-CF is a phase II, dose ranging, multicenter, double-blind, placebo controlled study to evaluate safety and effects of (R)-roscovitine in subjects with Cystic Fibrosis carrying 2 Cystic Fibrosis causing mutations with at least one F508del-CFTR mutation and chronically infected with Pseudomonas aeruginosa.

The aim of this study is to assess the safety of increasing doses of roscovitine administered orally for 4 cycles of 4 consecutive days (treatment "on") separated by a 3 days treatment free period (treatment "off") in 36 adult cystic fibrosis subjects.

These 36 patients will be allocated to 3 groups of 12 subjects who will be randomized in a 2:1 ratio (active drug to matching placebo). In each group, 8 patients will receive roscovitine (200 mg, 400 mg, 2 X 400 mg in group 1, 2 and 3, respectively) and 4 will receive a matching placebo. Treatment will be provided by oral administration of capsules. Each patient will receive the same treatment throughout the 28 day study.

This phase II trial will give some preliminary information about safety and hints of effects of a new experimental treatment. If the data suggest that a short term treatment with roscovitine provides a safe, effective and convenient approach for CF patients chronically infected with Pseudomonas aeruginosa, patients participating in this proof of concept trial will be offered to participate in further longer term studies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years of age on the date of informed consent;
* Diagnosed CF patients. Confirmed diagnosis of CF (Rosenstein and Cutting, 1998);
* Patients carrying 2 Cystic Fibrosis causing mutations with at least one F508del-CFTR mutation, genotype to be confirmed at screening;
* Forced expiratory volume at 1 second (FEV1) 40%
* Chronic lung Pseudomonas aeruginosa infection according to the definition from the French Consensus Conference;
* Able to understand and comply with all protocol requirements, restrictions and instructions and likely to complete the study as planned (as judged by the investigator);
* Provide written informed consent prior to the performance of any study-related procedure;

Exclusion Criteria:

* Acute upper or lower respiratory infection, pulmonary exacerbation or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before V2;
* Recent patient reported history of:

  * non recovered viral upper respiratory tract infection
  * solid organ or hematological transplantation
  * Burkholderia cepacia complex or Non Tuberculous Mycobacteria (NTM) respiratory tract infection;
* Undergone major surgery within 1 month prior to screening;
* Currently treated allergic broncho-pulmonary aspergillosis (ABPA);
* Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1C >8%;
* Hemoptysis more than 60 mL at any time within 4 weeks prior to first study drug administration (V2);
* History of any other comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject;
* Any other clinically significant conditions (not associated with the study indication) at Screening (V1) which might interfere with the assessment of this study;
* Any of the following abnormal laboratory values at screening:

  * Hemoglobin <10 g/dL
  * Abnormal liver function
  * Serum K+ <3,5 mmol/L
  * Abnormal renal function
* Any clinically significant laboratory abnormalities;
* Patients who have clinically significant impairment in cardiovascular function;
* Concomitant disease(s) that could prolong the QT interval;
* Patients with a history of alcohol or drug abuse in the past year;
* Patients with a history of noncompliance to medical regimens and patients or caregivers who are considered potentially unreliable;
* Use of one (or several) prohibited medications and/or food;
* Administration of any investigational drug within 30 days prior to Screening (V1) or 5 half-lives, whichever is longer;
* Use of systemic anti-pseudomonal antibiotics within 28 days prior to first study drug administration (V2). However use of inhaled anti-pseudomonal antibiotic treatment is allowed if initiated for more than 28 days;
* Use of loop diuretics within 7 days prior to first study drug administration (V2);
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Safety of increasing doses of Roscovitine | 3 months
  The primary objective of this study is to assess the safety of increasing doses of roscovitine administered orally for 4 cycles of 4 consecutive days (treatment "on") separated by a 3 days treatment free period (treatment "off") in adult CF subjects who carrying 2 Cystic Fibrosis causing mutations with at least F508del mutation

SECONDARY OUTCOMES:
Change in the concentration of Pseudomonas Aeruginosa | 3 months
  Change in the concentration (CFU/mL) of Pseudomonas aeruginosa in the sputum at each visit from V1 (Screening) up to V7 (Completion Visit).
PK parameters | 3 months
  PK parameters: Maximum Concentration (Cmax), Time to reach Cmax (Tmax), Area Under Curve (AUCt and AUCInf), Half-life (t1/2) for roscovitine and its M3 metabolite.
Pro- and anti-inflammatory cytokines | 3 months
  Monitoring the levels of pro- and anti-inflammatory cytokines, in particular: interleukin (IL)-17A, IL-5, IFN-γ, IL-1 receptor antagonist, IL-4, IL-6, IL-10, tumor necrosis factor-alpha, and IL-18 on V2, V3 and V7 (Completion Visit)
C-reactive protein | 3 months
  Change in C-reactive protein (CRP) at each visit from V1 (Screening) up to V7 (Completion)
Cystic Fibrosis Questionnaire-Revised | 3 months
  Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) at each visit from V1 up to V8 (Safety Follow-up)
Body Mass Index | 3 months
  Change in body mass index (BMI) at each visit from V1 (Screening) up to V7 (Completion Visit)
Forced expiratory volume in 1 second | 3 months
  Change in forced expiratory volume in 1 second (FEV1) at each visit from V1 (Screening) up to V7 (Completion Visit)
Sweat Chloride Concentration | 3 months
  Change in Sweat Chloride Concentration at V2, V3, V5 and V7 (Completion)
Nasal Potential Difference | 3 months
  Change in Nasal Potential Difference (NPD) at V1 (Screening) and V6 (for patients included in Paris Cochin CF Center)
Pain questionnaire | 3 months
  Evaluate of the pain and of the impact of the pain in patients with cystic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Gilles RAULT, MD, Principal Investigator — Centre de Pérharidy - Roscoff
Locations (11):
- France (11):
  - CHU de Nice - Hôpital Pasteur, Nice, France
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac, France
  - Centre de Ressources et de Compétences de la mucoviscidose, Reims, France
  - Centre Hospitalier Bretagne Atlantique, Vannes, France
  - CHR - Hôpital Calmette, Lille
  - CH Lyon Sud, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Cochin, Paris
  - Centre de Perharidy, Roscoff
  - Hôpital Larrey, Toulouse

REFERENCES:
- [Result] Meijer L, Hery-Arnaud G, Leven C, Nowak E, Hillion S, Renaudineau Y, Durieu I, Chiron R, Prevotat A, Fajac I, Hubert D, Murris-Espin M, Huge S, Danner-Boucher I, Ravoninjatovo B, Leroy S, Macey J, Urban T, Rault G, Mottier D, Berre RL. Safety and pharmacokinetics of Roscovitine (Seliciclib) in cystic fibrosis patients chronically infected with Pseudomonas aeruginosa, a randomized, placebo-controlled study. J Cyst Fibros. 2022 May;21(3):529-536. doi: 10.1016/j.jcf.2021.10.013. Epub 2021 Dec 24. PMID 34961705